CLINICAL TRIAL: NCT06724887
Title: Brain Health on College Campuses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Meadows Foundation (Unknown); Hoglund Foundation (Unknown)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Professor, Chief Director of UTD Center for BrainHealth, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-877
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Health Behavior; Life Style, Healthy
MeSH Terms: conditions — Health Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Health Training and Education (Experimental): Online and in-person training and education around brain-health strategies and lifestyle practices.
  Interventions: Behavioral: Brain Health Strategy Training and Education

INTERVENTIONS:
Behavioral: Brain Health Strategy Training and Education — Initial training strategies cover Strategic Memory Advanced Reasoning Tactics (SMART), and subsequent training extends the SMART principles to other life-applications such as stress management, sleep, and lifestyle. Virtual and in-person workshops will expand on topics such as stress management, sleep, resilience, and mental well-being, with an emphasis on how practicing and implementing brain healthy strategies can impact everyday life. For faculty/staff, we will also offer interactive workshops on how to create a brain healthy environment and classroom, including ways to implement and provide brain-healthy strategies and resources in their everyday operations involving students.

SUMMARY:
Center for BrainHealth is beginning a one-year pilot with local college campuses investigating the impact of (i) brain health assessment and training tools delivered through the online BrainHealth Platform and (ii) in-person educational brain health workshops delivered to college students and faculty/staff, with the overarching goal to better understand how to promote brain-healthier campuses (i.e., reflecting generally positive function across cognitive, social, emotional, and lifestyle domains). This initial study is intended to be a one-year pilot, with findings informing feasibility and efficacy as well as future, more extended and expanded study informing translation to other colleges/universities.

DETAILED DESCRIPTION:
ONLINE Procedures

Assessments (3 times over 9 months): BrainHealth Index - An online battery of cognitive measures and questionnaires. Periodic surveys to assess new research questions (as IRB approved) and to assess participant experience

Training, habits, resources (available over 9 months): Micro-learning video modules that include Strategic Memory Advanced Reasoning Tactics (SMART) and other trainings such as stress management, sleep, and lifestyle. The habit tool supports accountability and consistency of building new and personalized habits. Curated resources (articles, podcasts, videos) around the topic of brain health are also available.

Coaching Periodic access to group and one-on-one brain-health related virtual coaching sessions.

Link wearable data Participants have the option to link their wearable data with their data collected through the BrainHealth Platform

IN-PERSON Procedures

The investigators will offer in-person and/or virtual/hybrid educational sessions on a variety of high-interest topics such as stress management, sleep, resilience, and mental well-being, with an emphasis on how practicing and implementing brain healthy strategies can impact everyday life. For faculty/staff, the investigators will also offer interactive workshops on how to create a brain healthy environment and classroom, including ways to implement and provide brain-healthy strategies and resources in their everyday operations involving students (e.g., ways to enhance mental energy and focus in the classroom, brain-based approaches to promoting growth mindset and confidence, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* Either enrolled as a student and/or employed as staff/faculty at UTD or Dallas College
* Internet and device access
* Must be able to hear and read over the computer
* Fluent English speaker

Exclusion Criteria:

* Currently or previously enrolled in The BrainHealth Project (NCT04869111)
* Diagnosed neurodegenerative disease
* History of stroke, concussion, or brain injury that currently hinders participant from functioning at their prior level
* Diagnosed with autism spectrum disorder and not functioning independently

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
BrainHealth Index (BHI) | Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
  The investigators will assess change on a holistic measure of cognitive, social, well-being, and daily life health on the BrainHealth Index across multiple timepoints. (Min value = 16, Max value = 1032) (Higher score represents better outcome)

SECONDARY OUTCOMES:
Level of Real-Life Responsibilities Survey | Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
  A qualitative survey of with five sections: home, academic, job, extracurricular, and financial level of responsibilities. (Min value = 5, Max value = 15) (Higher score represents better outcome)_

OTHER OUTCOMES:
Grade Point Average (GPA) | Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
  A numerical representation of a student's overall academic performance (Min value = 0, Max value = 4.0)(Higher score represents better outcome)
Course Completion | Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
  Average course completion by student (Min value = 0, Max value = 100)(Higher score represents better outcome)
Program Retention and Completion | Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
  Average program retention and completion rates (Min value = 0, Max value = 100)(Higher score represents better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Cook, PhD, Principal Investigator — The University of Texas at Dallas
Locations (2):
- United States (2):
  - Dallas College, Dallas, Texas
  - University of Texas at Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman SB, Fratantoni JM, Robertson IH, D'Esposito M, Ling GSF, Zientz J, Vernon S, Venza E, Cook LG, Tate A, Spence JS. A Novel BrainHealth Index Prototype Improved by Telehealth-Delivered Training During COVID-19. Front Public Health. 2021 Mar 16;9:641754. doi: 10.3389/fpubh.2021.641754. eCollection 2021. PMID 33796498
- [Background] Zientz J, Spence JS, Chung SSE, Nanda U, Chapman SB. Exploring how brain health strategy training informs the future of work. Front Psychol. 2023 Sep 12;14:1175652. doi: 10.3389/fpsyg.2023.1175652. eCollection 2023. PMID 37771803
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Gamino JF, Chapman SB, Hull EL, Lyon GR. Effects of higher-order cognitive strategy training on gist-reasoning and fact-learning in adolescents. Front Psychol. 2010 Dec 9;1:188. doi: 10.3389/fpsyg.2010.00188. eCollection 2010. PMID 21833248